CLINICAL TRIAL: NCT06340282
Title: Effects of Immersive Virtual Reality and/or Multicomponent Physical Exercise on Cognitive and Functional Performance in Hospitalized Older Patients With Severe Functional Dependency: Study Protocol for a Randomized Clinical Trial
Brief Title: Immersive Virtual Reality and Physical Exercise on Cognitive and Functional Performance in Hospitalized Older Patients
Acronym: MOTOMED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MOTOMED
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Disability Physical; Cognition
Keywords: hospital-associated functional decline; cognitive stimulation; immersive virtual reality; multicomponent physical exercise; disability

STUDY DESIGN:
Intervention Model Description: This clinical randomized controlled trial will be conducted in the Acute Geriatric Unit of a tertiary hospital in Spain. A total of 212 acute patients will be enrolled according to the following criteria: age > 75, Barthel Index < 60, able to collaborate, expected length of stay > 5 days, absence of clinical instability and severe dementia (GDS 7) or other end-stage disease. Patients will be randomly assigned to a control group (CG) or any of the three intervention groups (IG): IVR, ME, or IVR + ME. The IVR group will watch ad-hoc videos showing Spanish regional landscapes and villages, approximately 4 minutes per day for three consecutive days. The ME group will undergo aerobic and strength exercise for progressive training of the upper and lower limbs. The IVR + ME group will do both cognitive and physical intervention. The primary outcomes will be cognitive and physical measures at discharge. Mood, quality of life, isometric strength, and acceptance of IVR will be also assessed.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Control group
- immersive virtual reality (Experimental): Patients use virtual reality
  Interventions: Device: Virtual reality
- multicomponent physical exercise intervention (Experimental): Individualized exercise intervention
  Interventions: Behavioral: multicomponent exercise
- Immersive virtual reality and multicomponent physical exercise intervention (Experimental): Both
  Interventions: Device: Virtual reality; Behavioral: multicomponent exercise

INTERVENTIONS:
Device: Virtual reality — Immersive virtual reality
  Arms: Immersive virtual reality and multicomponent physical exercise intervention; immersive virtual reality
Behavioral: multicomponent exercise — individualized exercise
  Arms: Immersive virtual reality and multicomponent physical exercise intervention; multicomponent physical exercise intervention

SUMMARY:
This study will be conducted in a hospital in Spain to investigate how a special intervention using immersive virtual reality technology can benefit hospitalized older adults with difficulties in their daily functionality.

The main objective of this study is to evaluate whether a cognitive stimulation intervention through immersive virtual reality, along with specific physical exercises, can improve the cognitive and physical function of hospitalized older patients. It is expected that this innovative intervention will have a positive impact on the quality of life of these patients.

Participants eligible for the study must be over 75 years old, have severe functional dependency upon hospital admission, and be willing to participate. Those with severe dementia or other terminal illnesses will be excluded.

Participants will be randomly assigned to one of four study groups: a control group without intervention and three intervention groups, including viewing Spanish landscapes through virtual reality, performing specific physical exercises, or a combination of both interventions.

At the end of the study, various aspects such as cognitive and physical function, mood, quality of life, muscle strength, and acceptance of virtual reality technology by patients will be evaluated.

This study aims to provide new insights into the care of hospitalized older adults and explore innovative ways to improve their well-being during their hospital stay

DETAILED DESCRIPTION:
This study will be conducted in a Spanish tertiary hospital to investigate the impact of a cognitive stimulation intervention through immersive virtual reality (IVR) on hospitalized older adults with severe functional dependency. The study will also examine the combined effect of a multicomponent exercise intervention (ME) with IVR. A total of 212 acute patients will be enrolled in the Acute Geriatric Unit of the hospital, meeting specific inclusion criteria related to age, stability in cardiopulmonary, respiratory, and neurological systems, expected length of stay, and ability to communicate and collaborate with the research team. Patients will be randomly assigned to a control group or one of three intervention groups: IVR, ME, or IVR + ME.

The interventions for the IVR and ME groups will involve watching 3D videos of Spanish landscapes and undergoing progressive upper and lower extremity exercises, respectively. The IVR + ME group will receive both interventions, while the control group will receive usual care. Primary outcome measures include cognitive tests, strength assessments, and balance and mobility evaluations. Secondary outcome measures include mood, quality of life, functional performance, delirium assessments, and length of hospital stay.

The study will take place in the Acute Geriatric Unit (AGU) of a tertiary hospital in Pamplona, Navarra, Spain, and will adhere to standard clinical trial guidelines. Eligibility criteria include medical inpatients admitted to the AGU between January 2024 and March 2025, with specific inclusion and exclusion criteria. The study aims to evaluate the impact of the interventions on cognitive and physical function among hospitalized older adults with severe functional dependency, with the goal of enhancing their well-being and care during hospitalization.

The research team anticipates that the interventions will positively influence cognitive function, physical performance, mood, quality of life, isometric strength, and acceptance of virtual reality technology among participants. The study's comprehensive approach encompasses various assessments to provide a holistic evaluation of the interventions' effectiveness in improving outcomes for hospitalized older adults with severe functional dependency.

Overall, this study represents a significant effort to understand how innovative interventions such as cognitive stimulation through IVR and multicomponent physical exercise could positively impact the health outcomes and quality of life of hospitalized older adults with severe functional dependency. The study's findings are expected to provide valuable insights for healthcare providers, researchers, and policymakers seeking to optimize care for this population.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 75 years Clinica Stability Expected length of stay ≥ 5 days Being able to communicate and collaborate with the research team

Exclusion Criteria:

Barthel Index score ≥ 60 at admission Refusal to sign the informed consent by the patient/legal guardian or inability to obtain it Life expectancy less than three months End-stage disease Severe level of major neurocognitive disorder (GDS 7)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE) | Baseline, day 3, at discharge and 1 month after discharge
  Cognitive evolution

SECONDARY OUTCOMES:
Isometric handgrip strength | Baseline, day 3, at discharge and 1 month after discharge
  Muscle strength measurement

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Martinez-Velilla Dr, PhD, Principal Investigator — Fundación Miguel Servet - Navarrabiomed
Locations (1):
- Hospital Universitario de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Yes
The plan to share anonymized data from a randomized clinical trial in response to reasonable requests focuses on ensuring confidentiality and protecting the privacy of participants. This plan includes fully anonymizing the data, creating a detailed data sharing protocol, establishing an independent data review committee, implementing a clear request procedure, requiring confidentiality agreements to be signed by requestors, and applying robust security measures to protect data integrity. The primary goal is to facilitate access to data to promote transparency and scientific advancement while ensuring respect for the privacy and confidentiality of clinical trial participants. It is important to note that data will be shared under reasonable requests.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the paper is published
Access Criteria: Any reasonable demand
URL: https://www.navarrabiomed.es/es

REFERENCES:
- [Result] Cuevas-Lara C, Saez de Asteasu ML, Ramirez-Velez R, Izquierdo M, Zambom-Ferraresi F, Antonanzas-Valencia C, Galbete A, Zambom-Ferraresi F, Martinez-Velilla N. Effects of game-based interventions on functional capacity in acutely hospitalised older adults: results of an open-label non-randomised clinical trial. Age Ageing. 2022 Jan 6;51(1):afab247. doi: 10.1093/ageing/afab247. PMID 35077558
- [Derived] de la Casa-Marin A, Zambom-Ferraresi F, Ferrara MC, Ollo-Martinez I, Galbete A, Gonzalez-Glaria B, Moral-Cuesta D, Marin-Epelde I, Chenhuichen C, Lorente-Escudero M, Molero-de-Avila R, Baztan AG, Zambom-Ferraresi F, Martinez-Velilla N. Effects of immersive virtual reality stimulation and/or multicomponent physical exercise on cognitive and functional performance in hospitalized older patients with severe functional dependency: study protocol for a randomized clinical trial. BMC Geriatr. 2024 Nov 8;24(1):924. doi: 10.1186/s12877-024-05516-x. PMID 39516806